CLINICAL TRIAL: NCT06194188
Title: A Phase 2 Clinical Study to Evaluate the Efficacy and Safety of CU-20401 for Injection in Moderate to Severe Contour Protuberance or Excessive Enrichment Due to Submental Fat (SMF) Accumulation
Brief Title: A Phase 2 Clinical Study of CU-20401
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CU-20401-203
Record Dates: First submitted 2023-11-30; First posted 2024-01-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Efficacy and Safety
Keywords: immunogenicity; SMF

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Group (Experimental): 0.06mg/ml/dose, the number of doses administered (no more than 36 doses) will be determined after the area has been assessed by the investigator based on the subject's submental fat accumulation
  Interventions: Drug: Subcutaneous injection of CU-20401
- High Dose Group (Experimental): 0.08 /ml/dose, the number of doses administered (no more than 36 doses) will be determined after the area has been assessed by the investigator based on the subject's submental fat accumulation
  Interventions: Drug: Subcutaneous injection of CU-20401
- Placebo group (Placebo Comparator): 0/ml/dose, the number of doses administered (no more than 36 doses) will be determined after the area has been assessed by the investigator based on the subject's submental fat accumulation
  Interventions: Drug: Subcutaneous injection of CU-20401

INTERVENTIONS:
Drug: Subcutaneous injection of CU-20401 — Reconstitute the product with 0.9% sodium chloride solution for injection, respectively, before use, for a single subcutaneous injection in the submental fat area.
  Other Names: cu-20401

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase Ⅱ clinical study to evaluate the efficacy, safety, and immunogenicity of CU-20401 for Injection in a population with moderate to severe contour elevation or over-fullness due to SMF accumulation.

DETAILED DESCRIPTION:
Eligible subjects were randomized in a 1: 1: 1 ratio to CU-20401 low dose group (0.06 mg/dose), CU-20401 high dose group (0.08 mg/dose), or placebo group using the severity of baseline clinician-reported SMF accumulation (score 2 or 3) as a stratification factor, and received a single subcutaneous injection of this group in the submental fat region on D1; return to the hospital for efficacy assessment on D29, D57, D85 or at early withdrawal; return to the hospital for safety assessment on D1, D8, D15, D29, D57, D85 or early withdrawal; immunogenicity samples were collected on D1, D8, D15, D29, D57, D85, or at early withdrawal (the study design is shown in the figure below).

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study contents, study process and possible adverse reactions, be able to complete the study in accordance with the protocol requirements, have reasonable expectations for the injection effect, and voluntarily sign the informed consent form;
2. Men or women aged 18 to 65 years (including boundary values) at the time of signing the ICF;
3. Body mass index (BMI) between 17 and 40 (kg/m2) at screening and baseline (including cut-off);
4. At screening and baseline, the investigator rated moderate to severe submental outline protrusion due to submental fat accumulation according to the clinician-reported Submental Fat Rating Scale (CR-SMFRS) , i.e., those with a score of 2 to 3 points; and the subject-reported Submental Fat Rating Scale (PR-SMFRS)rated the amount of submental fat as moderate/large/very large, i.e., those with a score of 2 to 4;
5. Subjects of childbearing potential (including males and females) have no pregnancy plans and voluntarily take effective contraceptive measures at screening and throughout the trial, and have no sperm or egg donation plans.

Exclusion Criteria:

1. Subjects who have received prior surgery, liposuction therapy, or injection of lipolytic drugs similar to the investigational drug (e.g., phosphatidylcholine, etc.) at the submental site;
2. Those who have received biomaterial fillings (e.g., hyaluronic acid, collagen, etc.) within 24 months prior to screening and at the neck or submental site before baseline;
3. Those who have received botulinum toxin injection within 3 months prior to screening and at the neck or submental site prior to baseline, or have received noninvasive skin tightening therapy;
4. Planned to undergo cosmetic procedures at the submental site during the study, including, but not limited to, dermal filling, surgical wrinkle removal, photoelectric therapy, water light needles, microneedles, chemical exfoliation, or scar removal surgery, etc.;
5. Enlargement of the submental area due to other causes of excess non-submental fat accumulation (e.g., goiter, lymphadenopathy, Madelong's disease, platysma protrusion at rest, etc.) or affect the investigator's assessment of submental fat;
6. Those with obvious scars, infections, cancerous or precancerous lesions and/or unresolved wounds, retrognathia, etc. in the chin and neck position, which may affect the evaluation results as assessed by the investigator;
7. According to the investigator's judgment, submental fat dissolution can cause submental skin relaxation (SMSLG) to be Grade 4 or have other anatomic features (e.g., bulging fat under the platysma, extreme skin relaxation of the neck or submental area, protrusion of the platysma band), resulting in unacceptable cosmetic results;
8. Subjects with a pre-existing tendency to scar hyperplasia or keloid may affect the efficacy assessment or subject safety after treatment as judged by the investigator;
9. Subjects with symptoms or associated diseases of dysphagia at screening and baseline;
10. Abnormal clinical laboratory tests (AST or ALT values above twice the upper limit of normal; serum creatinine above 1.5 times the upper limit of normal; triglycerides above 2 times the upper limit of normal) at screening and baseline; or other laboratory tests, vital signs, physical examination, electrocardiogram test results are abnormal and clinically significant, and the investigator considers it inappropriate to participate in this study;
11. Other acute or chronic diseases (including but not limited to cardiovascular and cerebrovascular, respiratory, endocrine, digestive, renal, liver, blood and lymphatic, immune, metabolic and skeletal, central nervous system or psychiatric disorders, etc.) at screening and baseline, which, as judged by the investigator, may increase the risk associated with the use of the investigational product, or may affect the interpretation of the study results, or fail to cooperate well with the study participant;
12. Hepatitis B surface antigen (HBsAg) positive, hepatitis C virus (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive, treponema pallidum antibody (TP-Ab) test positive at screening;
13. Clotting test results (prothrombin time, activated partial thromboplastin time) within 4 weeks prior to dosing indicate any clinically significant bleeding tendency (patients receiving antiplatelet, anticoagulant, acetylsalicylic acid therapy may be enrolled after a 7-day washout period);
14. Those who have used topical medications (e.g., glucocorticoids, tretinoin ointment) within 4 weeks prior to screening and in the prebaseline submental area, or are expected to require use in the submental area during the course of the study (up to 12 weeks after completion of injection);
15. Plan any surgery during the trial that may result in significant weight change (≥ 10%) or take any medication that may result in significant weight change (≥ 10%) (e.g. systemic corticosteroids, bariatric medications, bariatric surgery);
16. Donation of blood or massive blood loss (≥ 400 mL) within 3 months prior to screening and prior to baseline;
17. History of needle sickness and blood sickness;
18. History of drug abuse within 6 months prior to screening and prior to baseline, or drug use within 3 months prior to screening and prior to baseline;
19. Allergic constitution, or history of allergy to collagenase or components of the study drug or its excipients;
20. Received collagenase treatment within 6 months prior to screening and prior to baseline;
21. Those who have participated in any drug or medical device clinical trials within 3 months before screening and before baseline or within 1 month before screening and before baseline;
22. Lactating and pregnant women;
23. Those who cannot undergo magnetic resonance imaging (MRI) (e.g., with a pacemaker/electronic stimulator, an insulin pump, a cochlear implant, or stainless steel metal implanted in the body, etc.);
24. Other conditions judged by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
change in both CR-SMFRS score and PR-SMFRS score at the same time | Day 29
  at least 1 point change in both clinician-reported Submental Fat Rating Scale (CR-SMFRS) score and subject-reported Submental Fat Rating Scale (PR-SMFRS) score 爱at the same time.
  CR-SMFRS score ,0=None,1=Minor,2=Moderate,3=Serious,4=very severe. PR-SMFRS score,0=None,1=very little,2=a little,3=a few，4=a lot

SECONDARY OUTCOMES:
Proportion of subjects with at least 1 point change in CR-SMFRS score and PR-SMFRS score | Day 57/ Day 85
  Proportion of subjects with at least 1 point change in clinician-reported Submental Fat Rating Scale (CR-SMFRS) score and subject-reported Submental Fat Rating Scale (PR-SMFRS) score.
  CR-SMFRS score ,0=None,1=Minor,2=Moderate,3=Serious,4=very severe. PR-SMFRS score,0=None,1=very little,2=a little,3=a few，4=a lot
Proportion of subjects with at least 2 points change in CR-SMFRS score and PR-SMFRS score | Day 29/Day 57/Day 85
  Proportion of subjects with at least 2 points change in clinician-reported Submental Fat Rating Scale (CR-SMFRS) score and subject-reported Submental Fat Rating Scale (PR-SMFRS) score.
  CR-SMFRS score ,0=None,1=Minor,2=Moderate,3=Serious,4=very severe. PR-SMFRS score,0=None,1=very little,2=a little,3=a few，4=a lot
change from baseline in CR-SMFRS score | Day 29/Day 57/Day 85
  change from baseline in clinician-reported Submental Fat Rating Scale (CR-SMFRS) score，0=None,1=Minor,2=Moderate,3=Serious,4=very severe
change from baseline in PR-SMFRS score | Day 29/Day 57/Day 85
  change from baseline insubject-reported Submental Fat Rating Scale (PR-SMFRS) score. ,0=None,1=very little,2=a little,3=a few,4=a lot
Change from baseline in the total score of PR-SMFIS | Day 29/Day 57/Day 85
  Change from baseline in the total score of Submental Fat Impact Scale (PR-SMFIS) ,1=euphoria in the subject's mood ,2=distress,3=cares about，4=embarrassed about,5= look old,6=look overweight
Proportion of subjects with at least a 10% reduction from baseline in submental fat volume using MRI | Day 29/Day 85
  Proportion of subjects with at least a 10% reduction from baseline in submental fat volume using MRI
MRI was used to examine the change from baseline in submental fat volume | Day 29/Day 85
  MRI was used to examine the change from baseline in submental fat volume
MRI was used to examine the change from baseline in submental fat thickness | Day 29/Day 85
  MRI was used to examine the change from baseline in submental fat thickness
Change from baseline in Submental Skin Relaxity Scale (SMSLG) | Day 85
  Change from baseline in SMSLG score,1=None，2=Minor，3=Moderate，4=Serious

CONTACTS AND LOCATIONS:
Overall Officials: byron Zhu, MD, Study Chair — CMO
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China